CLINICAL TRIAL: NCT02980419
Title: Erticality Perception - Effects of Prolonged Roll-tilt in Healthy Human Subjects
Brief Title: Effects of Prolonged Roll-tilt in Healthy Human Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: post_tilt_study
Record Dates: First submitted 2016-11-16; First posted 2016-12-02 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Adaptation Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention arm (Experimental): In each participant the investigators will assess verticality perception in whole-body upright position by use of the SVV, the SPV and the SHV after static roll-tilt at ±90deg over 5min. Measurements will be obtained on a motor-driven turntable and two different roll-tilt positions will be applied (±90°). A visual line (SVV), a rod (SHV) or the turntable itself will be adjusted to indicate perceived direction of vertical. A total of three measuring sessions, each lasting about 60 minutes are scheduled.
  Interventions: Behavioral: presentation of visual and vestibular stimuli

INTERVENTIONS:
Behavioral: presentation of visual and vestibular stimuli — In each participant the investigators will assess verticality perception in whole-body upright position by use of the SVV, the SPV and the SHV after static roll-tilt at ±90deg over 5min. Measurements will be obtained on a motor-driven turntable and two different roll-tilt positions will be applied (±90°). A visual line (SVV), a rod (SHV) or the turntable itself will be adjusted to indicate perceived direction of vertical. A total of three measuring sessions, each lasting about 60 minutes are scheduled.

SUMMARY:
The long-term goal of this research is to advance the investigators knowledge of how the brain combines the information of multiple sensory systems coding for spatial oriention and how adaptation to vestibular imbalance influences spatial orientation. In healthy human subjects verticality perception is accurate while upright. After prolonged roll-tilt, humans show a systematic bias in perceived direction towards the previous roll-tilted position (so-called "post-tilt bias"). This effect could either be related to adaptation to the roll-tilted position (shifting the "null" position) or it could be related to changes in torsional eye position due to prolonged static roll-tilt (ocular counter-roll). While in the first case a post-tilt bias is predicted independently of the experimental paradigm used, the second hypothesis predicts a post-tilt bias only if retinal cues are integrated. In order to evaluate these hypotheses, the investigators will assess perceived vertical using both vision-dependent and vision-independent paradigms.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-65 years
* informed consent
* absence of exclusion criteria

Exclusion Criteria:

* peripheral-vestibular deficit
* disturbed consciousness
* history of sensory deficits
* visual field deficits
* other neurological or systemic disorder which can cause dementia or cognitive dysfunction
* intake of antidepressants, sedatives, or neuroleptics
* pregnancy, unless excluded by a negative pregnancy test
* known neck pain or status post neck trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
adjustment errors of the subjective visual/haptic/postural vertical in upright position after prolonged whole-body roll-tilt positions. | 10 minutes (i.e. short-term adaptation)
  the accuracy and precision of visual vertical adjustments after prolonged roll tilt are quantified.

SECONDARY OUTCOMES:
changes in adjustment errors of the subjective visual vertical when providing an additional optokinetic stimulus | 10 minutes (i.e. short-term adaptation)
  This is the same as in outcome 1, but an additional visual (optokinetic) stimulus is added
changes in adjustment errors of the subjective haptic vertical when providing an additional optokinetic stimulus | 10 minutes (i.e. short-term adaptation)
  This is the same as in outcome 1, but an additional visual (optokinetic) stimulus is added
changes in adjustment errors of the subjective postural vertical when providing an additional optokinetic stimulus | 10 minutes (i.e. short-term adaptation)
  This is the same as in outcome 1, but an additional visual (optokinetic) stimulus is added

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Dept. of Neurology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No